CLINICAL TRIAL: NCT07338045
Title: The Effects of Eight-Week Baduanjin Exercise on Chronic Low Back Pain and Disability Among Office Workers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Professor, School of Medical Sciences, Universiti Sains Malaysia, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/25030299
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain; Baduanjin
Keywords: Office Workers; Non-pharmacological Intervention
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is a parallel-group randomized controlled trial with two arms: the Baduanjin intervention group and the control group. Participants were randomly assigned to one of the two groups. The intervention lasted for 8 weeks, during which the Baduanjin group received structured exercise training, while the control group did not receive any structured exercise intervention. After completion of post-intervention data collection, participants in the control group were offered access to the Baduanjin program as part of an ethical follow-up measure.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was blinded to group assignment during all assessment procedures. Participants were assessed using standardized tools (VAS, CODI, Berg Balance Scale...) by a trained evaluator who was unaware of the participant's group allocation. All assessments were conducted in a neutral environment without any reference to intervention status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin group (Experimental): The Baduanjin group convened at 5:00 p.m. on a daily basis for a period of one hour, five days a week, for a total of eight weeks. The intervention period involved a total of 40 exercises. The Baduanjin exercise was overseen by two senior coaches with a minimum of five years' experience in physical education.The training programme for the eight-duanjin exercise was based on the Fitness Qigong - Baduanjin, a publication by the State General Administration of Sport, which includes ten postures (including the beginning and ending postures) (Li et al., 2015).
  Interventions: Behavioral: Baduanjin Exercise Program
- Control group (Active Comparator): During the 8-week intervention period, participants in the control group will not receive any structured exercise intervention, including the Eight-Week Baduanjin Exercise Program or other physical therapy programs. They will continue with their usual daily activities without additional guidance related to low back pain management. After completion of the post-intervention data collection, participants in the control group will be offered access to the Eight-Week Baduanjin Exercise Program as a form of ethical follow-up, conducted under the supervision of a trained instructor.
  Interventions: Other: Usual Care / No Structured Exercise

INTERVENTIONS:
Behavioral: Baduanjin Exercise Program — A traditional Chinese qigong-based exercise program involving eight gentle movements designed to promote circulation, strengthen muscles, and improve balance. Participants will attend supervised sessions five times per week for 8 weeks, each lasting 45 minutes.
  Arms: Baduanjin group
Other: Usual Care / No Structured Exercise — Participants will continue with their regular daily activities without receiving any structured exercise intervention or specific guidance related to low back pain management during the 8-week study period. They will be provided with information about the Baduanjin Exercise Program after the completion of all data collection, as part of an ethical follow-up measure.
  Arms: Control group

SUMMARY:
Office workers often suffer from chronic low back pain due to long hours of sitting and poor posture. This study will test whether Baduanjin-a gentle, traditional Chinese exercise-can help reduce pain and improve physical function in office staff with long-standing back pain. Thirty participants will be randomly assigned to either practice Baduanjin for eight weeks or receive no special intervention. Researchers will measure changes in pain levels, movement ability, balance, posture, and daily functioning before and after the program. Baduanjin is a safe, low-cost, and easy-to-learn exercise that could be widely used in community health settings as a non-drug therapy for back pain.

DETAILED DESCRIPTION:
The modern office environment has led to increased sedentary behavior and poor postures among office workers, contributing significantly to chronic low back pain (LBP) and associated functional impairments. This condition not only reduces work productivity and quality of life but also increases healthcare costs and societal burden.

This randomized controlled trial aims to evaluate the effects of an eight-week Baduanjin exercise program on pain intensity, physical function, and disability in office workers with chronic LBP. Thirty eligible participants will be randomly allocated to either the Baduanjin group or a control group. The Baduanjin group will attend supervised Baduanjin training sessions three times per week for eight weeks, while the control group will maintain their usual routine without any specific intervention.

Outcome assessments will be conducted at baseline and immediately after the 8-week intervention. Primary outcomes include: (1) pain severity measured by the Visual Analog Scale (VAS); (2) joint mobility assessed using the Joint Mobility Scale; (3) balance function evaluated via the Berg Balance Scale; (4) postural risk analyzed by the Rapid Entire Body Assessment (REBA); and (5) lumbar spine dysfunction determined by the Chinese version of the Oswestry Disability Index (CODI).

Data will be analyzed using SPSS version 17.0. Continuous variables will be presented as mean ± standard deviation. A two-way repeated-measures ANOVA will be used to examine the interaction effects between group (Baduanjin vs. control) and time (pre- vs. post-intervention). A p-value < 0.05 will be considered statistically significant.

Findings from this study may support the integration of Baduanjin into primary healthcare and community-based rehabilitation programs as a safe, simple, and effective non-pharmacological intervention for chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

-

This study specifically targets office workers diagnosed with mechanical (or non-specific) chronic low back pain, which refers to persistent low back pain without a specific identifiable pathological cause such as disc herniation, spinal stenosis, or inflammatory diseases. Mechanical low back pain is the most common form of chronic low back pain among sedentary populations, particularly office workers, and is primarily attributed to musculoskeletal imbalances, poor posture, and prolonged sitting.Participants were included in the study if they met the following criteria:

1. Age and Occupational Requirements: Office workers between the ages of 20 and 55 years with at least two years of continuous employment.
2. History of Chronic Low Back Pain: Presence of persistent or recurrent low back pain localized below the costal margin and above the inferior gluteal folds, with a duration of more than three months.
3. Pain Intensity Assessment: A pain score exceeding 40 mm on a 100 mm Visual Analogue Scale (VAS), indicating a moderate level of pain.
4. Clinical Diagnosis Confirmation: Participants must be diagnosed with mechanical (non-specific) chronic low back pain by orthopaedic sports medicine specialists from the First Affiliated Hospital of Xi'an Jiaotong University. All participants will be required to submit their annual full-body medical examination report provided by the university between May 30 and July 30 each year. The Principal Investigator will collect these reports in advance and arrange for orthopaedic sports medicine specialists from the affiliated hospital to conduct an on-site screening at Xi'an Jiaotong University City College. During this process, specialists will review participants' medical history, evaluate physical symptoms, and consider available imaging reports (e.g., X-rays or MRI scans if previously conducted) to confirm the absence of specific spinal pathologies such as disc herniation or spinal stenosis. These specialists are experts in diagnosing and managing musculoskeletal conditions related to physical activity and sports, ensuring accurate assessment and classification of participants' chronic low back pain. Their involvement guarantees both clinical validity and safety in participant selection.
5. Cognitive and Physical Function: Normal cognitive function, adequate communication and interaction skills, and the physical ability to perform the basic movements of Baduanjin exercise. Participants must also have voluntarily provided written informed consent and agreed to comply with all study procedures throughout the research period.
6. Employment Status: Staff members currently employed at Xi'an Jiaotong University City College. This criterion ensures that the study population consists exclusively of sedentary office workers within the university setting, enhancing homogeneity and relevance to the target demographic.

Exclusion Criteria:

-

Subjects are excluded from this study if they:

1. Those with other spinal pathologies such as lumbar fractures, lumbar disc herniation, spondylolisthesis, intravertebral occupancy, lumbar spinal stenosis, and severe osteoporosis. These conditions may interfere with the interpretation of outcomes related to chronic low back pain of non-specific origin, and could also affect the safety or effectiveness of the Baduanjin exercise intervention.
2. Persons with contraindications such as leukaemia, thrombocytopenia and other diseases with bleeding tendency, acute infectious diseases and oncological diseases. These systemic illnesses may affect participant safety or confound the results, and are therefore not included in the target population of office workers with chronic low back pain.
3. Suffering from diseases of liver and kidney function, serious cardiac disorders, and other diseases affecting the study. The presence of these comorbidities could influence the ability of participants to safely complete the Baduanjin exercise program, and thus they are excluded to ensure homogeneity among the target group of individuals with chronic low back pain.
4. Women who are pregnant. Pregnancy-related changes in posture and musculoskeletal loading can affect low back pain symptoms and response to exercise, which may confound the study findings.
5. Subjects who do not agree to sign the informed consent form. All participants will be required to submit their annual full-body medical examination report provided by the university between May 30 and July 30 each year. The Principal Investigator will collect these reports in advance and arrange for orthopaedic sports medicine specialists from the affiliated hospital to conduct an on-site screening at Xi'an Jiaotong University City College. During this process, the specialists will review all relevant medical findings, including imaging results, laboratory tests, and physician notes, to identify any conditions that meet the exclusion criteria. Participants found to have spinal pathologies, systemic illnesses, or other comorbidities that may affect safety, intervention effectiveness, or study outcomes will be excluded from the study. These exclusion criteria are designed to ensure that the final sample consists exclusively of individuals with mechanical (non-specific) low back pain, thereby enhancing the homogeneity of the study population and minimizing confounding factors in evaluating the effects of Baduanjin exercise.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, 8 weeks post-intervention
  A 100-mm horizontal line where participants mark their perceived level of low back pain intensity, with 0 mm indicating no pain and 100 mm indicating worst possible pain. The distance from 0 to the mark is measured in millimeters and used as the score.

SECONDARY OUTCOMES:
Joint Mobility Scale | Baseline, 8 weeks post-intervention
  The Joint Mobility Scale is used to assess the functional status of the spine and surrounding structures. Joint mobility in all directions of the lumbar region was measured using a joint mobility measuring tape.
Berg Balance Scale | Baseline, 8 weeks post-intervention
  A standardized test assessing balance function through 14 tasks such as sitting to standing, turning, and reaching. Each task is scored from 0 to 4, with a total score ranging from 0 to 56. Higher scores indicate better balance.
Rapid Entire Body Assessment (REBA) | Baseline, 8 weeks post-intervention
  An ergonomic risk assessment tool that evaluates posture and movement during work tasks to identify potential musculoskeletal risks. It provides a risk score based on body position and force requirements.
Chinese version of the Lumbar Spine Dysfunction Index (CODI) | Baseline, 8 weeks post-intervention
  A validated questionnaire assessing functional limitations and disability related to low back pain. It includes items on daily activities, work, and social functioning. Higher scores indicate greater dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Xi'an Jiaotong University City College, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qi Y, Zhuang M, Liang R, Shaharudin S. The effect of traditional Chinese exercises on low Back pain and disability in middle-aged and older adults: A systematic review. Prev Med Rep. 2025 Apr 14;54:103072. doi: 10.1016/j.pmedr.2025.103072. eCollection 2025 Jun. PMID 40290641